CLINICAL TRIAL: NCT00001861
Title: Screening Study for the Evaluation and Diagnosis of Potential Research Subjects With Nystagmus or Strabismus
Brief Title: Screening for Studies on Nystagmus and Strabismus
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990035; 99-EI-0035
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Nystagmus; Strabismus
Keywords: Eye Movements; Amblyopia; Orthoptics; Lazy Eye; Eye Development; Nystagmus; Strabismus; Screening Protocol; Eye Movement Disorders
MeSH Terms: conditions — Nystagmus, Pathologic; Strabismus; Amblyopia; Ocular Motility Disorders

SUMMARY:
This screening protocol is designed to help recruitment patients for National Eye Institute (NEI) studies on nystagmus and strabismus. Patients must meet specific requirements of a research study, and this protocol serves as a first step for admitting patients to an appropriate program.

Candidates will undergo a medical history, physical examination, eye examination and blood test. The eye examination includes measurement of eye pressure and dilation of the pupils to fully examine the lens, vitreous and retina. Specialized tests will be done only if needed to determine eligibility for a nystagmus or strabismus study. These include routine laboratory tests, non-invasive imaging, questionnaires, and other standard tests. If needed, a test called oculography may be done to record eye movements. There are two procedures for recording and documenting these movements. In the infrared system, the patient wears a pair of glasses or goggles and looks at a red light while the head is kept steady. In the search coil system, the eye is numbed with anesthetic eye drops and a soft contact lens is placed on the eye. Then the patient looks at a red light while the head is held still. Each oculography session lasts 20 to 30 minutes. Photographs of the eye may be taken.

When the screening is completed, patients will be informed of their options to participate in a study. Patients who are ineligible for a current study will be informed of alternative treatments or options. No treatment is offered under this protocol.

DETAILED DESCRIPTION:
This protocol is designed for the screening of patients with either diagnosed or undiagnosed conditions, and serves as a first step for individuals who may be eligible and wish to participate in National Eye Institute (NEI) clinical research studies.

Each individual will be thoroughly evaluated during the screening process to determine if they are suitable candidates for inclusion in any of the NEI ongoing studies. The screening evaluation will include past and current medical histories, and an appropriate physical examination. Other routine diagnostic procedures and tests may also be completed in order to help determine a subject's eligibility. These tests and procedures are of minimal risk. Once the screening process is completed and their eligibility assessed, the subjects will be informed of their options to participate in one or more of the current clinical research studies. If no appropriate protocol is identified, recommendations for other treatment options may be given to the individual, their primary doctor or referring physician.

ELIGIBILITY:
* INCLUSION CRITERIA

Inclusion and exclusion criteria vary with the particular protocol for which a patient is being screened.

In addition to those diagnoses currently under study, subjects with unusual, interesting, or unknown conditions that require the establishment of a diagnosis may be eligible for inclusion in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 1999-01-29; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Miura K, Hertle RW, FitzGibbon EJ, Optican LM. Effects of tenotomy surgery on congenital nystagmus waveforms in adult patients. Part I. Wavelet spectral analysis. Vision Res. 2003 Oct;43(22):2345-56. doi: 10.1016/s0042-6989(03)00409-7. PMID 12962991